CLINICAL TRIAL: NCT06737861
Title: Effects of Buerger Exercises With Whole Body Vibration on Pain, Balance and Lower Limb Perfusion in Patients With Diabetic Peripheral Neuropathy
Brief Title: Buerger Exercises With Whole Body Vibration in Diabetic Peripheral Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/0262 Malaika Shahid
Record Dates: First submitted 2024-12-12; First posted 2024-12-17 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Diabetic Peripheral Neuropathic Pain; Balance Changes; Ankle Brachial Index
Keywords: Buerger Exercises; Whole Body Vibration Therapy; Diabetic peripheral neuropathy

STUDY DESIGN:
Intervention Model Description: interventional study model for this study is a parallel-group randomized controlled trial (RCT). This model involves two distinct groups:
  Intervention Group: Participants receive both Buerger exercises and Whole Body Vibration (WBV) therapy.
  Control Group: Participants receive only Buerger exercises without WBV therapy. Each participant is assigned randomly to one of these groups, ensuring that comparisons between the combined therapy and single therapy are unbiased. This parallel structure means each group undergoes its specific intervention throughout the study period without crossover to the other group's intervention. This approach helps assess the distinct and combined effects of the two therapies on pain, balance, and lower limb perfusion in patients with diabetic peripheral neuropathy.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): Buerger exercises and Whole Body Vibration (WBV) exercise group
  Interventions: Other: Group A
- Group B (Active Comparator): Buerger exercises group
  Interventions: Other: Group B

INTERVENTIONS:
Other: Group A — Participants will perform Buerger exercises three times daily, with each session including three cycles. Additionally, they will receive Whole Body Vibration therapy at a frequency of 25 Hz, three times per week. Each WBV session will last 12 minutes, divided into four 3-minute bouts, aiming to improve pain, balance, and lower limb circulation in diabetic peripheral neuropathy patients.
  Other Names: Buerger exercises with Whole Body Vibration
  Arms: Group A
Other: Group B — Participants will perform Buerger exercises three times daily, with each session consisting of three cycles. This exercise regimen is aimed at assessing its effectiveness on pain, balance, and circulation in diabetic peripheral neuropathy patients, serving as a comparison to the combined intervention with WBV therapy.
  Other Names: Buerger exercises
  Arms: Group B

SUMMARY:
The goal of this clinical trial is to determine if a combined intervention of Buerger exercises and whole-body vibration therapy can improve pain, circulation, and balance in adults with diabetic peripheral neuropathy.

Participants will:

Perform Buerger exercises three times daily in both groups. Receive whole-body vibration therapy three times per week (intervention group only).

Complete assessments at baseline, the 4th, 8th, 12th weeks, and a follow-up at the 16th week.

Outcome measures include pain rating, ankle-brachial index, balance scale, and timed mobility test. Statistical analyses will assess within-group and between-group effects based on data distribution.

DETAILED DESCRIPTION:
This study, titled "Effects of Buerger Exercises with Whole Body Vibration on Pain, Balance, and Lower Limb Perfusion in Patients with Diabetic Peripheral Neuropathy," aims to assess the combined effectiveness of Buerger exercises and Whole-Body Vibration (WBV) therapy in addressing diabetic peripheral neuropathy (DPN). DPN is a common complication of diabetes mellitus, affecting roughly 50% of diabetic individuals globally and leading to sensory impairments, pain, mobility issues, and an elevated risk for severe foot complications. In Pakistan, where a large population suffers from diabetes, there is an urgent need for effective interventions for DPN. Existing research has shown that Buerger exercises alone are beneficial in improving lower limb circulation, the ankle-brachial index, and capillary refill time, while also reducing neuropathy risk by promoting blood circulation to the lower limbs. Separately, WBV therapy has demonstrated improvements in sensory perception, neuropathy scores, balance, and quality of life, as well as enhanced muscle strength and reflex responses through motor unit activation. Despite this evidence, the combined effect of these two interventions has not been studied extensively, creating a research gap regarding their potential synergistic benefits. This study seeks to fill that gap by evaluating outcomes in pain, balance, and circulation among DPN patients receiving both interventions, with the hypothesis that the combination may be more effective than Buerger exercises alone.

This randomized controlled trial (RCT) will be conducted at Civil Hospital Sialkot and Social Security Hospital Sialkot and is expected to last ten months. Participants, aged 50-70 and diagnosed with DPN, will be randomly assigned to two groups: an intervention group that receives both Buerger exercises and WBV therapy, and a control group performing only Buerger exercises. WBV therapy sessions will occur three times weekly at a frequency of 25 Hz, each lasting 12 minutes with a protocol of four 3-minute bouts. The Buerger exercises will be performed daily by both groups, with three cycles per session and three sessions per day. Outcomes will be measured using the Numeric Pain Rating Scale (NPRS) for pain assessment, the Ankle-Brachial Index (ABI) for lower limb perfusion, the Berg Balance Scale (BBS) for balance, and the Timed Up and Go Test (TUGT) for functional mobility. Data collection will take place at baseline, the 4th, 8th, and 12th weeks, and there will be a follow-up at the 16th week to determine if the benefits are sustained.

The study will recruit participants who meet specific inclusion criteria, such as having an HbA1c level higher than 6.7 mmol/L and MNSI scores indicating DPN, while excluding those with severe pain, cardiovascular conditions, deep vein thrombosis, or advanced diabetes complications like diabetic foot. A single-blinded approach will be used to ensure that outcome assessors are not aware of the participant's group allocation. Data will be analyzed using SPSS-27, with normality checks via Kolmogorov-Smirnov and Shapiro-Wilk tests. If data is normally distributed, within-group comparisons will use Repeated Measures ANOVA and between-group comparisons will use one-way ANOVA; if data is not normally distributed, the Mann-Whitney U test will be used for between-group comparisons and the Friedman test for within-group comparisons.

This study is significant in that it will address a clinical gap by evaluating the combined impact of Buerger exercises and WBV therapy on pain, balance, and circulation in individuals with DPN. If successful, it could offer a more effective treatment option to improve quality of life and functionality in this patient population. The study timeline includes major milestones such as title approval, synopsis defense, data collection, analysis, and a final report, all aimed at completing the study within ten months after approval. Ethical considerations have been meticulously planned, with informed consent processes in both English and Urdu to ensure participants' understanding and voluntary involvement. This research has the potential to provide meaningful insights into a novel intervention strategy for DPN management, which could be beneficial in both clinical practice and future research applications.

ELIGIBILITY:
Inclusion criteria:

* Participants with both genders male and female will be included in the study.
* The Age limit for the participants will be 50-70 years.
* Patients diagnosed with diabetes from last 5 Years.
* The participants with Hb1Ac higher than 6.7mmol/L.
* Patients diagnosed with diabetic peripheral neuropathy with scores ≥ 4 on Michigan Neuropathy Screening Instrument (MNSI).
* Patients with Ankle Brachial Index < 1-1.2mmHg.
* Those patients who were able to participate in exercise interventions.

Exclusion criteria:

* The patients with Numeric Pain Rating Scale values greater than 4.
* Patients with severe cardiovascular or musculoskeletal conditions contraindicating exercise.
* Patients with serious mental problems or inability to communicate.
* Patients with Deep venous thrombosis.
* Patients with Diabetic foot ulcers or foot gangrene.
* Patients having serious complications of diabetes, such as amputation and patients who are unable to complete the entire program.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2024-12-20 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Ankle Brachial Index (ABI) | Assessment at baseline after, 4th, 8th, 12th and 16th week
  The ABI is a non-invasive measure of lower limb perfusion, calculated as the ratio of ankle systolic blood pressure to brachial systolic blood pressure. An improvement in ABI suggests better blood circulation, which is a key outcome for assessing the intervention's effect on lower limb vascular health.

SECONDARY OUTCOMES:
Numeric Pain rating Scale (NPRS) | Assessment at baseline after, 4th, 8th, 12th and 16th week
  NPRS is an 11-point scale ranging from 0 (no pain) to 10 (worst pain imaginable), used to measure the intensity of pain experienced by participants. This self-reported scale helps quantify pain levels and gauge the effectiveness of the intervention on pain reduction.
Mini-Balance Evaluation Systems Test (Mini-BESTest) | Assessment at baseline after, 4th, 8th, 12th and 16th week
  MiniBESTest is 14 items, each scored on a 3-point scale (0 = severe impairment, 2 = normal), with a maximum score of 28.
  Covers four balance domains:
  Anticipatory postural adjustments (e.g., sit-to-stand, rise on toes) Reactive postural control (compensatory stepping responses) Sensory orientation (balance under altered sensory conditions) Dynamic gait (dual-task walking, pivot turns, speed changes) Lower scores indicate poorer balance and higher fall risk. A cut-off score of ≤19/28 is often used to identify individuals at risk of falls.

OTHER OUTCOMES:
Timed Up and Go Test (TUGT) | Assessment at baseline, after 4th, 8th, 12th and 16th weeks
  TUGT is a functional mobility test where participants are timed as they stand from a seated position, walk 3 meters, turn around, walk back, and sit down. The test assesses mobility and balance, with faster completion times indicating better mobility and balance.

CONTACTS AND LOCATIONS:
Overall Officials: Aruba Saeed, PhD, Principal Investigator — Riphah International University
Locations (1):
- Social Security Hospital in Sialkot, Sialkot, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akbari NJ, Naimi SS. The effect of exercise therapy on balance in patients with diabetic peripheral neuropathy: a systematic review. J Diabetes Metab Disord. 2022 Jul 4;21(2):1861-1871. doi: 10.1007/s40200-022-01077-1. eCollection 2022 Dec. PMID 36404857
- [Background] Gomes-Neto M, de Sa-Caputo DDC, Paineiras-Domingos LL, Brandao AA, Neves MF, Marin PJ, Sanudo B, Bernardo-Filho M. Effects of Whole-Body Vibration in Older Adult Patients With Type 2 Diabetes Mellitus: A Systematic Review and Meta-Analysis. Can J Diabetes. 2019 Oct;43(7):524-529.e2. doi: 10.1016/j.jcjd.2019.03.008. Epub 2019 Mar 27. PMID 31104903
- [Background] Ahmad AM, Mohammed AA, Khalifa WA, Ali HM, Abdel-Aziz A. Effect of Buerger-Allen exercise on wound healing in patients with diabetic foot ulcers: a randomised controlled trial. J Wound Care. 2024 Apr 2;33(Sup4a):xci-xcviii. doi: 10.12968/jowc.2024.33.Sup4a.xci. PMID 38588058
- [Background] Kessler NJ, Lockard MM, Fischer J. Whole body vibration improves symptoms of diabetic peripheral neuropathy. J Bodyw Mov Ther. 2020 Apr;24(2):1-3. doi: 10.1016/j.jbmt.2020.01.004. Epub 2020 Feb 11. PMID 32507132
- [Background] Jamal A, Ahmad I, Ahamed N, Azharuddin M, Alam F, Hussain ME. Whole body vibration showed beneficial effect on pain, balance measures and quality of life in painful diabetic peripheral neuropathy: a randomized controlled trial. J Diabetes Metab Disord. 2019 Dec 21;19(1):61-69. doi: 10.1007/s40200-019-00476-1. eCollection 2020 Jun. PMID 32550157
- [Background] Radhika J, Poomalai G, Nalini S, Revathi R. Effectiveness of Buerger-Allen Exercise on Lower Extremity Perfusion and Peripheral Neuropathy Symptoms among Patients with Diabetes Mellitus. Iran J Nurs Midwifery Res. 2020 Jun 17;25(4):291-295. doi: 10.4103/ijnmr.IJNMR_63_19. eCollection 2020 Jul-Aug. PMID 33014740